CLINICAL TRIAL: NCT02046863
Title: DBS-Expert: Automated Deep Brain Stimulation Programming Using Functional Mapping - Phase I
Brief Title: Pilot Study for Automated Deep Brain Stimulation Programming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1R43NS081902-01 (NIH); 1R43NS081902 (NIH)
Record Dates: First submitted 2013-12-05; First posted 2014-01-28 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-08

CONDITIONS: Parkinson's Disease; Tremor; Bradykinesia
Keywords: Parkinson's disease; Tremor; Bradykinesia; Deep brain stimulation; Kinesia
MeSH Terms: conditions — Parkinson Disease; Tremor; Hypokinesia

ARMS (1):
- Automated Programming (Experimental): Subjects will have DBS settings changed as guided by prototype DBS-Expert software. Tremor, bradykinesia, and dyskinesia will be assessed at each DBS setting.
  Interventions: Device: Automated Programming

INTERVENTIONS:
Device: Automated Programming — Prototype DBS-Expert software will be used to guide a clinician through DBS programming.

SUMMARY:
The clinical utility of deep brain stimulation (DBS) for the treatment of movement disorders such as Parkinson's disease has been well established; however, there is a great disparity in outcomes among DBS recipients due to varied postoperative management, particularly concerning the choosing of an optimal set of programming parameters from the thousands of possible combinations. This study will evaluate the use of motion sensor based assessments to develop a functional map and algorithms to automatically determine a set of programming parameters that maximize symptomatic benefits while minimizing side effects and battery consumption.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease
* Implanted deep brain stimulation system awaiting initial programming session

Exclusion Criteria:

* Subjects with significant psychiatric illness or dementia
* Significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin A Heldman, PhD, Principal Investigator — Great Lakes NeuroTechnologies
Locations (1):
- University of Cincinnati Department of Neurology, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Heldman DA, Pulliam CL, Urrea Mendoza E, Gartner M, Giuffrida JP, Montgomery EB Jr, Espay AJ, Revilla FJ. Computer-Guided Deep Brain Stimulation Programming for Parkinson's Disease. Neuromodulation. 2016 Feb;19(2):127-32. doi: 10.1111/ner.12372. Epub 2015 Dec 1. PMID 26621764

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Automated Programming
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Automated Programming
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 62 [54 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Kinesia HomeView Symptom Ratings After Guided DBS Programming
Description: Symptoms were first assessed with the implanted pulse generator (IPG) turned off for at least 30 minutes to allow the after-effects of stimulation to wear off (baseline). Symptoms were measured again with the IPG turned on at a setting that both minimized the average severity of tremor and bradykinesia and minimized side effects. The Kinesia score rated symptom severity (0, normal; 4, most severe) in four categories: tremor, finger tapping speed, finger tapping amplitude, and finger tapping rhythm. Scores for the four motor symptoms were averaged and converted to percent change from baseline.
Time Frame: Within two days of standard clinical DBS programming session
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Automated Programming
Number analyzed (Participants) | 7
Percentage change | -35.7 (37.8)

ADVERSE EVENTS:
Arm/Group | Automated Programming
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less